CLINICAL TRIAL: NCT02471222
Title: Safety and Efficacy of ADS-5102 (Amantadine HCl) Extended Release Capsules in Patients With Multiple Sclerosis and Walking Impairment
Brief Title: Safety and Efficacy of ADS-5102 in Patients With Multiple Sclerosis and Walking Impairment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Adamas Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADS-AMT-MS201
Record Dates: First submitted 2015-06-11; First posted 2015-06-15 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Walking Impairment; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ADS-5102 (amantadine HCl extended release) (Experimental)
  Interventions: Drug: ADS-5102
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ADS-5102 — Oral capsules to be administered once daily at bedtime for 4 weeks
  Other Names: amantadine HCl extended release
  Arms: ADS-5102 (amantadine HCl extended release)
Other: Placebo — Oral capsules to be administered once daily at bedtime for 4 weeks
  Arms: Placebo

SUMMARY:
This is a multi-center, randomized, double-blind, placebo-controlled, 2-arm, parallel group study of ADS-5102 extended release (ER) capsules, an investigational formulation of amantadine, dosed once daily at bedtime for the treatment of walking impairment in MS. ADS-5102 is designed to be administered once daily at bed time, ADS-5102 achieves higher plasma amantadine concentrations in the early morning, sustained throughout the afternoon, and lower concentrations in the evening when patients are sleeping. ADS-5102 is designed to deliver its primary treatment effect during the day, and potentially reduce the adverse events of immediate-release amantadine when the patient is asleep.

ELIGIBILITY:
Inclusion Criteria:

* Signed a current IRB-approved informed consent form;
* Male or female subjects between 18 and 70 years of age, inclusive;
* Confirmed diagnosis of Multiple Sclerosis according to the 2010 Revised McDonald criteria;
* On a stable regimen of medications taken specifically to treat MS for at least 30 days prior to screening, and willing to continue the same doses and regimens for the duration of study participation;
* Stable physical activity level for at least 30 days prior to screening and willing to continue without change for the duration of study participation;
* Maximum EDSS score during screening of 6.5;
* Sufficient ambulatory ability to complete two trials of the Timed 25 Foot Walk (T25FW) at the screening visit;
* A score on each completed screening T25FW test between 8 and 45 seconds, inclusive;
* Any other current and allowed prescription/non-prescription medications and/or nutritional supplements taken regularly must have been at a stable dose and regimen for at least 30 days prior to screening, and subject must be willing to continue the same doses and regimens during study participation;
* If taking an antidepressant, must be on a stable dose for at least 60 days prior to screening.

Exclusion Criteria:

* History of seizures within 2 years prior to screening;
* Clinically significant MS relapse with onset less than 30 days prior to screening;
* Presence of vertigo or other vestibular dysfunction that might compromise ability to safely perform the T25FW;
* Received physical therapy within 30 days prior to screening;
* Received systemic steroids within 30 days prior to screening;
* Received dalfampridine, methylphenidate, modafinil, armodafinil, amantadine, and/or any product containing amphetamines, or any treatment specifically for fatigue or to improve walking within 30 days prior to screening;
* Received any botulinum toxin containing product used as antispasmodic agent within 3 months prior to screening;
* History of clinically significant hallucinations due to an MS medication or other/unknown cause, within 2 years prior to screening;
* History of Bipolar Disorder or Psychosis, regardless of treatment;
* Presence of cognitive impairment sufficient, in the opinion of the investigator, to affect the subject's ability to complete study assessments, or which would not be in the subject's best interest to participate in the study;
* History of stroke or TIA within 2 years prior to screening;
* History of cancer within 5 years;
* Presence of untreated angle closure glaucoma;
* If female, is pregnant or lactating;
* If a sexually active female, is not surgically sterile or at least 2 years post-menopausal, or does not agree to utilize a highly effective hormonal method of contraception (an IUD, or vasectomized male partner is also acceptable), in combination with a barrier method, from screening through at least 4 weeks after the completion of study treatment;
* Treatment with an investigational drug or device within 30 days prior to screening;
* Treatment with an investigational biologic within 6 months prior to screening;
* Current participation in another clinical trial;
* Planned elective surgery during study participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-05; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Safety of ADS-5102 assessed by adverse events, safety-related study drug discontinuations, vital signs, and safety laboratory test | Up to 4 weeks

SECONDARY OUTCOMES:
Timed 25 Foot Walk | Up to 4 weeks
Timed Up and go | Up to 4 weeks
2 Minute Walk Test | Up to 4 weeks
MS Walking Scale-12 | Up to 4 weeks

OTHER OUTCOMES:
Fatigue Scale for Motor and Cognitive Functions | Up to 4 weeks
Beck's Depression Inventory-2 | Up to 4 weeks
Brief International Cognitive Assessment for MS | Up to 4 weeks

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Phoenix, Arizona
  - Aurora, Colorado
  - Sarasota, Florida
  - Atlanta, Georgia
  - Northbrook, Illinois
  - Rochester, Minnesota
  - Lincoln, Nebraska
  - Albuquerque, New Mexico
  - Patchogue, New York
  - Raleigh, North Carolina
  - Cleveland, Ohio
  - Oklahoma City, Oklahoma
  - Franklin, Tennessee
  - Dallas, Texas
  - Kirkland, Washington